CLINICAL TRIAL: NCT04929626
Title: Comparison of Doses of Nebulized Magnesium Sulphate as an Adjuvant Treatment With Salbutamol in Children With Status Asthmaticus
Brief Title: Different Doses of Nebulized Magnesium Sulphate in Status Asthmaticus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr.Rabia Asif, Principal investigator, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Doses of Nebulized MgSO4
Record Dates: First submitted 2021-05-10; First posted 2021-06-18 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Status Asthmaticus
Keywords: asthma; nebulized; magnesium sulphate
MeSH Terms: conditions — Status Asthmaticus; Asthma | interventions — Magnesium Sulfate; Albuterol

STUDY DESIGN:
Intervention Model Description: Eligible patients were divided in two groups. In group A, patients received 3 back-to-back nebulization with Ventolin solution only using nebulizer machine and face mask after every 20 minutes for 60 minutes. In group B, patients were divided into 3 subgroups and each subgroup received both Ventolin and MgSO4 with three different doses after every 20 minutes for 60 minutes
Who Masked: Participant, Care Provider
Masking Description: The principal investigator was aware of the intervention being provided. Others were masked including the participant and care provider.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebulized Ventolin (Active Comparator): Nebulized Ventolin will given to 1st group after every 20 min for 1 hour
  Interventions: Drug: Ventolin
- Nebulized Magnesium Sulphate + Ventolin (Experimental): Dose of Nebulized Magnesium sulphate will vary in 3 subgroups.
  Interventions: Drug: Magnesium Sulfate 500 mg/ml+ ventolin

INTERVENTIONS:
Drug: Magnesium Sulfate 500 mg/ml+ ventolin — 3 doses of magnesium sulphate i.e; 250mg(0.5ml), 500mg(1ml), 750mg(1.5ml) will be used in nebulized form
  Other Names: MgSO4
  Arms: Nebulized Magnesium Sulphate + Ventolin
Drug: Ventolin — it will be given to control group in nebulized form after every 20 min in 1st hour
  Other Names: Salbutamol
  Arms: Nebulized Ventolin

SUMMARY:
In this study investigators will use magnesium sulphate in the nebulized form in children between 2 and 12 years of age as an acute reliever for acute severe asthma. Aim of this study is to determine that whether adding low (250mg), intermediate (500mg), and high doses (750mg) of magnesium sulphate in the 1st hour of treatment has any difference in the improvement of clinical condition of the patient and length of hospital stay. There will be total 108 patients having 2 groups. 1st group will receive only Ventolin while 2nd group will be given Ventolin and Magnesium sulphate.

DETAILED DESCRIPTION:
This randomized clinical trial will include 126 patients after taking informed consent who will meet the eligibility criteria. Patients will be randomly distributed in 2 groups on alternate basis as computerized generated number. Improvement will be assessed in terms of clinical condition i.e., Heart Rate, Respiratory Rate, blood pressure, pattern of breathing oxygen saturation and Pediatric Respiratory Assessment Measure (PRAM) score at start of treatment and then afterwards at 20 min interval up to 1 hour and then at 2nd hour and then after every 6 hours for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 2 to 12 years of age.
2. Children with the diagnosis of asthma having a pram score of more than 4.
3. Children with reactive airways

Exclusion Criteria:

1. Critically ill children who require intubation or mechanical ventilation.
2. Having hypersensitivity or allergy to MgSO4.
3. with history of chronic lung impairment.
4. Whose parents are not giving informed consent for participation in research.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Respiratory Assessment Measure (PRAM) score from the baseline | 20, 40, 60, 120, 360, 720, 1080, 1440 minutes after commencement of treatment
  The outcome measure was the response to treatment in terms of change in Pediatric Respiratory Assessment Measure (PRAM) score from the baseline, i.e; suprasternal indrawing, scalene retractions, wheezing, air entry, oxygen saturation on room air. Change in PRAM score means decrease in score i.e; mild (0-4), moderate (5-8), severe(9-12), impending respiratory failure (12+).
Change from baseline Suprasternal indrawing | 20, 40, 60, 120, 360, 720, 1080, 1440 minutes after commencement of treatment
  Absent (0) , Present (2)
Change from baseline Scalene retractions | 20, 40, 60, 120, 360, 720, 1080, 1440 minutes after commencement of treatment
  Absent (0) , Present (2)
Change from baseline Wheezing | 20, 40, 60, 120, 360, 720, 1080, 1440 minutes after commencement of treatment
  Absent (0), Expiratory only (1), Inspiratory and expiratory (2) Audible without (3) stethoscope/silent chest with minimal air entry
Change from baseline Air entry | 20, 40, 60, 120, 360, 720, 1080, 1440 minutes after commencement of treatment
  Normal (0), Decreased at bases (1), Widespread decrease (2), Absent/minimal (3)
Change from baseline Oxygen saturation on room air | 20, 40, 60, 120, 360, 720, 1080, 1440 minutes after commencement of treatment
  >93% (0), 90%-93% (1) or <90% (2)

SECONDARY OUTCOMES:
Hospital stay | 24 hours
  curtailment in the length of hospital stay
Hospital stay | 48 hours
  curtailment in the length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Asif, MBBS, PGT, Principal Investigator — Ziauddin Hospital
Locations (1):
- Rabia Asif, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alansari K, Ahmed W, Davidson BL, Alamri M, Zakaria I, Alrifaai M. Nebulized magnesium for moderate and severe pediatric asthma: A randomized trial. Pediatr Pulmonol. 2015 Dec;50(12):1191-9. doi: 10.1002/ppul.23158. Epub 2015 Feb 4. PMID 25652104
- [Background] Mustafa J, Iqbal SMJ, Azhar IA, Sultan MA. Nebulized magnesium sulphate as an adjunct therapy in the management of children presenting with acute exacerbation of asthma. Pakistan J Med Heal Sci. 2018;12(2):554-5.
- [Background] Daengsuwan T, Watanatham S. A comparative pilot study of the efficacy and safety of nebulized magnesium sulfate and intravenous magnesium sulfate in children with severe acute asthma. Asian Pac J Allergy Immunol. 2017 Jun;35(2):108-112. doi: 10.12932/AP0780. PMID 27996280
- [Background] Turker S, Dogru M, Yildiz F, Yilmaz SB. The effect of nebulised magnesium sulphate in the management of childhood moderate asthma exacerbations as adjuvant treatment. Allergol Immunopathol (Madr). 2017 Mar-Apr;45(2):115-120. doi: 10.1016/j.aller.2016.10.003. Epub 2017 Jan 31. PMID 28153353
- [Background] Sarhan HA, El-Garhy OH, Ali MA, Youssef NA. The efficacy of nebulized magnesium sulfate alone and in combination with salbutamol in acute asthma. Drug Des Devel Ther. 2016 Jun 9;10:1927-33. doi: 10.2147/DDDT.S103147. eCollection 2016. PMID 27354766
- [Background] Schuh S, Sweeney J, Freedman SB, Coates AL, Johnson DW, Thompson G, Gravel J, Ducharme FM, Zemek R, Plint AC, Beer D, Klassen T, Curtis S, Black K, Nicksy D, Willan AR; Pediatric Emergency Research Canada Group. Magnesium nebulization utilization in management of pediatric asthma (MagNUM PA) trial: study protocol for a randomized controlled trial. Trials. 2016 May 24;17(1):261. doi: 10.1186/s13063-015-1151-x. PMID 27220675
- [Background] Kew KM, Kirtchuk L, Michell CI. Intravenous magnesium sulfate for treating adults with acute asthma in the emergency department. Cochrane Database Syst Rev. 2014 May 28;2014(5):CD010909. doi: 10.1002/14651858.CD010909.pub2. PMID 24865567
- [Background] Akter T, Islam N, Hoque MA, Khanam S, Saha BK. Original Article Nebulization by Isotonic Magnesium Sulphate Solution with Salbutamol Provide Early and Better Response as Compared to Conventional Approach ( Salbutamol Plus Normal Saline ) in Acute Exacerbation of Asthma in Children . 2014;9(2):61-7.
- [Background] Powell CV, Kolamunnage-Dona R, Lowe J, Boland A, Petrou S, Doull I, Hood K, Williamson PR; MAGNETIC study group. MAGNEsium Trial In Children (MAGNETIC): a randomised, placebo-controlled trial and economic evaluation of nebulised magnesium sulphate in acute severe asthma in children. Health Technol Assess. 2013 Oct;17(45):v-vi, 1-216. doi: 10.3310/hta17450. PMID 24144222
- [Background] Hendaus MA, Jomha FA, Alhammadi AH. Is ketamine a lifesaving agent in childhood acute severe asthma? Ther Clin Risk Manag. 2016 Feb 22;12:273-9. doi: 10.2147/TCRM.S100389. eCollection 2016. PMID 26955277
- [Background] Dexheimer JW, Abramo TJ, Arnold DH, Johnson KB, Shyr Y, Ye F, Fan KH, Patel N, Aronsky D. An asthma management system in a pediatric emergency department. Int J Med Inform. 2013 Apr;82(4):230-8. doi: 10.1016/j.ijmedinf.2012.11.006. Epub 2012 Dec 4. PMID 23218449
- [Background] Kumar A. Effectiveness of Nebulized Magnesium Sulphate as an Adjuvant Therapy (With Salbutamol) in the Management of Acute Asthma. Pakistan J Med Dent. 2020;9(02):39-44.
- [Background] Reddel HK, Bateman ED, Becker A, Boulet LP, Cruz AA, Drazen JM, Haahtela T, Hurd SS, Inoue H, de Jongste JC, Lemanske RF Jr, Levy ML, O'Byrne PM, Paggiaro P, Pedersen SE, Pizzichini E, Soto-Quiroz M, Szefler SJ, Wong GW, FitzGerald JM. A summary of the new GINA strategy: a roadmap to asthma control. Eur Respir J. 2015 Sep;46(3):622-39. doi: 10.1183/13993003.00853-2015. Epub 2015 Jul 23. PMID 26206872
- [Background] Al-Shamrani A, Al-Harbi AS, Bagais K, Alenazi A, Alqwaiee M. Management of asthma exacerbation in the emergency departments. Int J Pediatr Adolesc Med. 2019 Jun;6(2):61-67. doi: 10.1016/j.ijpam.2019.02.001. Epub 2019 Mar 15. No abstract available. PMID 31388549
- [Background] Rehder KJ. Adjunct Therapies for Refractory Status Asthmaticus in Children. Respir Care. 2017 Jun;62(6):849-865. doi: 10.4187/respcare.05174. PMID 28546381
- [Background] Indinnimeo L, Chiappini E, Miraglia Del Giudice M; Italian Panel for the management of acute asthma attack in children Roberto Bernardini. Guideline on management of the acute asthma attack in children by Italian Society of Pediatrics. Ital J Pediatr. 2018 Apr 6;44(1):46. doi: 10.1186/s13052-018-0481-1. PMID 29625590
- [Background] Schuh S, Macias C, Freedman SB, Plint AC, Zorc JJ, Bajaj L, Black KJ, Johnson DW, Boutis K. North American practice patterns of intravenous magnesium therapy in severe acute asthma in children. Acad Emerg Med. 2010 Nov;17(11):1189-96. doi: 10.1111/j.1553-2712.2010.00913.x. PMID 21175517
- [Background] Goodacre S, Cohen J, Bradburn M, Gray A, Benger J, Coats T; 3Mg Research Team. Intravenous or nebulised magnesium sulphate versus standard therapy for severe acute asthma (3Mg trial): a double-blind, randomised controlled trial. Lancet Respir Med. 2013 Jun;1(4):293-300. doi: 10.1016/S2213-2600(13)70070-5. Epub 2013 May 17. PMID 24429154
- [Background] Ibrahim Z, Modawi FS, Almehaid AM, Alshenaifi NA, Albahouth ZI. REVIEW OF THE RECENT UPDATES REGARDING ACUTE ASTHMA EXACERBATION MANAGEMENT IN CHILDREN : A SIMPLE LITERATURE REVIEW Corresponding author : 2019;06(01):850-5
- [Background] Petrou S, Boland A, Khan K, Powell C, Kolamunnage-Dona R, Lowe J, Doull I, Hood K, Williamson P. Economic evaluation of nebulized magnesium sulphate in acute severe asthma in children. Int J Technol Assess Health Care. 2014 Oct;30(4):354-60. doi: 10.1017/S0266462314000440. Epub 2014 Nov 14. PMID 25394502
- [Background] Shein SL, Speicher RH, Filho JO, Gaston B, Rotta AT. Contemporary treatment of children with critical and near-fatal asthma. Rev Bras Ter Intensiva. 2016 Jun;28(2):167-78. doi: 10.5935/0103-507X.20160020. PMID 27305039
- [Derived] Asif R, Rais H, Bai P, Aziz R. Comparison of doses of Nebulized Magnesium sulphate as an adjuvant treatment with salbutamol in children with Status Asthmaticus. Pak J Med Sci. 2024 May-Jun;40(5):927-932. doi: 10.12669/pjms.40.5.7682. PMID 38827880
- See also: North American practice patterns of intravenous magnesium therapy in severe acute asthma in children — https://pubmed.ncbi.nlm.nih.gov/21175517/
- See also: Nebulized magnesium for moderate and severe pediatric asthma: A randomized trial — https://pubmed.ncbi.nlm.nih.gov/25652104/
- See also: A comparative pilot study of the efficacy and safety of nebulized magnesium sulfate and intravenous magnesium sulfate in children with severe acute asthma — https://pubmed.ncbi.nlm.nih.gov/27996280/
- See also: The effect of nebulised magnesium sulphate in the management of childhood moderate asthma exacerbations as adjuvant treatment — https://pubmed.ncbi.nlm.nih.gov/28153353/
- See also: The efficacy of nebulized magnesium sulfate alone and in combination with salbutamol in acute asthma — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4907636/
- See also: Magnesium nebulization utilization in management of pediatric asthma (MagNUM PA) trial: study protocol for a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/27220675/
- See also: Intravenous magnesium sulfate for treating adults with acute asthma in the emergency department — https://pubmed.ncbi.nlm.nih.gov/24865567/
- See also: Nebulization by Isotonic Magnesium Sulphate Solution with Salbutamol Provide Early and Better Response as Compared to Conventional Approach (Salbutamol Plus Normal Saline) in Acute Exacerbation of Asthma in Children — https://www.banglajol.info/index.php/FMCJ/article/view/25675
- See also: MAGNEsium Trial In Children (MAGNETIC): a randomised, placebo-controlled trial and economic evaluation of nebulised magnesium sulphate in acute severe asthma in children — https://pubmed.ncbi.nlm.nih.gov/24144222/
- See also: Is ketamine a lifesaving agent in childhood acute severe asthma? — https://pubmed.ncbi.nlm.nih.gov/26955277/
- See also: An asthma management system in a pediatric emergency department — https://pubmed.ncbi.nlm.nih.gov/23218449/
- See also: A summary of the new Global Initiative for Asthma (GINA) strategy: a roadmap to asthma control — https://pubmed.ncbi.nlm.nih.gov/26206872/
- See also: Management of asthma exacerbation in the emergency departments — https://pubmed.ncbi.nlm.nih.gov/31388549/
- See also: Adjunct Therapies for Refractory Status Asthmaticus in Children — https://pubmed.ncbi.nlm.nih.gov/28546381/
- See also: Guideline on management of the acute asthma attack in children by Italian Society of Pediatrics — https://pubmed.ncbi.nlm.nih.gov/29625590/
- See also: Intravenous or nebulised magnesium sulphate versus standard therapy for severe acute asthma (3Mg trial): a double-blind, randomised controlled trial — https://pubmed.ncbi.nlm.nih.gov/24429154/
- See also: Economic evaluation of nebulized magnesium sulphate in acute severe asthma in children — https://pubmed.ncbi.nlm.nih.gov/25394502/
- See also: Contemporary treatment of children with critical and near-fatal asthma — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4943055/